CLINICAL TRIAL: NCT00327015
Title: A Multicenter, Randomized, Double-Blind Active-Controlled, Phase 3 Trial to Evaluate the Efficacy and Safety of Saxagliptin in Combination With Metformin IR as Initial Therapy Compared to Saxagliptin Monotherapy and to Metformin IR Monotherapy in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control
Brief Title: A Phase 3 Study of BMS-477118 in Combination With Metformin in Subjects With Type 2 Diabetes Who Are Not Controlled With Diet and Exercise
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV181-039
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Results first posted 2009-09-25 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — saxagliptin; Metformin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Saxagliptin and Metformin (A) (Experimental): PLUS open-label pioglitazone (as needed as rescue medication)
  Interventions: Drug: Saxagliptin; Drug: Metformin; Drug: pioglitazone
- Saxagliptin and Metformin (B) (Experimental): PLUS open-label pioglitazone (as needed as rescue medication)
  Interventions: Drug: Saxagliptin; Drug: Metformin; Drug: pioglitazone
- Saxagliptin and Placebo (C) (Experimental): PLUS open-label pioglitazone (as needed as rescue medication)
  Interventions: Drug: Saxagliptin; Drug: Placebo; Drug: pioglitazone
- Metformin and Placebo (D) (Active Comparator): PLUS open-label pioglitazone (as needed as rescue medication)
  Interventions: Drug: Metformin; Drug: Placebo; Drug: pioglitazone

INTERVENTIONS:
Drug: Saxagliptin — Coated Tablets, Oral, 10 mg, Daily (6 months ST, 12 months LT)
  Other Names: BMS-477118
  Arms: Saxagliptin and Metformin (A); Saxagliptin and Placebo (C)
Drug: Saxagliptin — Coated tablets, PO, 5 mg, Daily (6 months ST, 12 months LT)
  Other Names: BMS-477118
  Arms: Saxagliptin and Metformin (B)
Drug: Metformin — Coated tablets, Oral, 500 mg, Daily (6 months ST, 12 months LT)
  Arms: Metformin and Placebo (D); Saxagliptin and Metformin (A); Saxagliptin and Metformin (B)
Drug: Placebo — Coated tablets, Oral, 0 mg, Daily (6 months ST, 12 months LT)
  Arms: Metformin and Placebo (D); Saxagliptin and Placebo (C)
Drug: pioglitazone — Tablets, Oral, 15-45 mg, as needed (12 months LT)

SUMMARY:
The purpose of this trial is to understand if adding saxagliptin to metformin therapy is safe and works better than taking either saxagliptin or metformin alone

DETAILED DESCRIPTION:
All subjects will participate in a lead-in period, and qualifying subjects will continue into a short-term randomized treatment period. Subjects who complete the short-term period will be eligible to enter the long term extension period. Also, subjects in the short-term period who have an elevated blood sugar that requires additional medication for blood sugar control will be eligible to enter the long-term treatment extension period where they will receive pioglitazone (rescue medication) added onto their blinded study medication

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Inadequate blood sugar control
* No current treatment with other medications to lower blood sugar

Exclusion Criteria:

* Major heart, liver or kidney problems
* Pregnant or breast feeding

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1306 (Actual)
Dates: Start 2006-05; Primary Completion 2007-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (159):
- United States (47):
  - East Bay Clinical Trial Center, Concord, California
  - Encompass Clinical Research, Encinitas, California
  - Community Clinical Trials, Orange, California
  - Coastal Biomedical Research Inc, Santa Monica, California
  - Encompass Clinical Research, Spring Valley, California
  - St. Joseph'S Medical Associates, Stockton, California
  - Clinical Therapeutics Corporation, Coral Gables, Florida
  - Florida Research Network, Llc, Gainesville, Florida
  - Fpa Clinical Research, Kissimmee, Florida
  - Emerald Coast Research Group, Marianna, Florida
  - Baptist Diabetes Associates, Miami, Florida
  - Middle Georgia Drug Study Center, Llc, Perry, Georgia
  - Cedar Crosse Research Center, Chicago, Illinois
  - Adviso Medical Research, Llc, Chicago, Illinois
  - Deerbrook Medical Associates, Vernon Hills, Illinois
  - Physicians Research Group, Indianapolis, Indiana
  - Professional Network Research Of Kansas, Wichita, Kansas
  - Medical Arts Research Collaborative, Llc, Excelsior Springs, Missouri
  - Nevada Alliance Against Diabetes, North Las Vegas, Nevada
  - Metrolina Medical Research, Charlotte, North Carolina
  - Durham Internal Medicine Assoc., Durham, North Carolina
  - Down East Medical Associates, Morehead City, North Carolina
  - Midwest Regional Research, Inc., Bellbrook, Ohio
  - Massillon Family Practice, Massillon, Ohio
  - Your Diabetes Endocrine Nutrition Group, Mentor, Ohio
  - Newark Physician Associates, Newark, Ohio
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Safe Harbor Clinical Research, East Providence, Rhode Island
  - Internal Medicine Of Greer, Greer, South Carolina
  - Middle Tennessee Clinical Research, Fayetteville, Tennessee
  - Frontier Clinical Research, Llc., Memphis, Tennessee
  - Capital Medical Clinic, Llp, Austin, Texas
  - Endocrine Associates, Houston, Texas
  - Advances In Health,Inc, Houston, Texas
  - Juno Research, Llc, Houston, Texas
  - Non Invasive Cardiovascular Pa, Houston, Texas
  - Tiena Health Research, Irving, Texas
  - Diabetes Center Of The Southwest, Midland, Texas
  - Hill Country Medical Associates, New Braunfels, Texas
  - Pearland Primary Care Associates, Llp, Pearland, Texas
  - Med-Cure Primary Care Physicians, Rosenberg, Texas
  - Gsa Research, San Antonio, Texas
  - Covenant Clinical Research, Pa, San Antonio, Texas
  - S.A.M. Clinical Research Center, San Antonio, Texas
  - Seven Corners Medical Research Center, Falls Church, Virginia
  - Salem Va Medical Ctr Research & Devlopment, Salem, Virginia
  - Physicians Clinic Of Spokane, Spokane, Washington
- Argentina (15):
  - Local Institution, Belgrano, Buenos Aires
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Chacabuco, Buenos Aires
  - Local Institution, La Plata, Buenos Aires
  - Local Institution, Morón, Buenos Aires
  - Local Institution, San Martín, Buenos Aires
  - Local Institution, San Pedro, Buenos Aires
  - Local Institution, Zárate, Buenos Aires
  - Local Institution, Mendoza, Mendoza Province
  - Local Institution, Salta, Salta Province
  - Local Institution, San Juan, San Juan Province
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, Lanus Este, Tucumán Province
  - Local Institution, Buenos Aires
- Brazil (8):
  - Local Institution, Fortaleza, Ceará
  - Local Institution, Goiânia, Goiás
  - Local Institution, Belém, Pará
  - Local Institution, Recife, Pernambuco
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Campinas, São Paulo
  - Local Institution, Marília, São Paulo
  - Local Institution, São Paulo, São Paulo
- Germany (13):
  - Local Institution, Aschaffenburg
  - Local Institution, Bad
  - Local Institution, Dresden
  - Local Institution, Duisburg
  - Local Institution, Heidelberg
  - Local Institution, Künzing
  - Local Institution, Ludwigshafen
  - Local Institution, Magdeburg
  - Local Institution, Mainz
  - Local Institution, Mannheim
  - Local Institution, Saarbrücken
  - Local Institution, Vellmar
  - Local Institution, Wangen
- Hungary (5):
  - Local Institution, Eger
  - Local Institution, Érd
  - Local Institution, Gyula
  - Local Institution, Szentes
  - Local Institution, Szigetvár
- India (12):
  - Local Institution, Panjagutta, Hyderabad, Andhra Pradesh
  - Local Institution, Vasanth Nagar, Bangalore
  - Local Institution, Bangalore, Karnataka
  - Local Institution, Pune, Maharashtra
  - Local Institution, Kandivili West, Mumbai
  - Local Institution, Sarita Vihar, New Delhi
  - Local Institution, Chennai, Tamil Nadu
  - Local Institution, Bangalore
  - Local Institution, Chennai
  - Local Institution, Haryāna
  - Local Institution, Rajasthan
  - Local Institution, Vellore, Tamilnadu
- Italy (5):
  - Local Institution, Catania
  - Local Institution, Genova
  - Local Institution, Milan
  - Local Institution, Perugia
  - Local Institution, Ravenna
- Mexico (7):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Cuernavaca, Morelos
  - Local Institution, Garza García, Nuevo León
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Mérida, Yucatán
- Philippines (6):
  - Local Institution, Cebu City
  - Local Institution, Iloilo City
  - Local Institution, Manila
  - Local Institution, Marikina City
  - Local Institution, Pasig
  - Local Institution, Quezon City
- Poland (9):
  - Local Institution, Gniewkowo
  - Local Institution, Gorzów Wielkopolski
  - Local Institution, Izabelin
  - Local Institution, Krakow
  - Local Institution, Lublin
  - Local Institution, Michalow-Regionow
  - Local Institution, Warsaw
  - Local Institution, Wroclaw
  - Local Institution, Zabrze
- Puerto Rico (4):
  - Local Institution, Carolina
  - Local Institution, Ponce
  - Local Institution, Rio Pieoras
  - Local Institution, San Juan
- Russia (21):
  - Local Institution, Kemerovo, Russia
  - Local Institution, Moscow, Russia
  - Local Institution, Nizhny Novgorod, Russia
  - Local Institution, Izhevsk
  - Local Institution, Kirov
  - Local Institution, Krasnodar
  - Local Institution, Kursk
  - Local Institution, Moscow
  - Local Institution, Nizhny Novgorod
  - Local Institution, Novosibirsk
  - Local Institution, Perm
  - Local Institution, Rostov-on-Don
  - Local Institution, Saint Peterburg
  - Local Institution, Saint Petersburg
  - Local Institution, Saratov
  - Local Institution, Smolensk
  - Local Institution, Tuymen
  - Local Institution, Vladimir
  - Local Institution, Volgograd
  - Local Institution, Yaroslaval
  - Local Institution, Yaroslavl
- Ukraine (7):
  - Local Institution, Dniepropetrovsk
  - Local Institution, Kharkiv
  - Local Institution, Kyiv
  - Local Institution, Lutsk
  - Local Institution, Lviv
  - Local Institution, Odesa
  - Local Institution, Ternopil

REFERENCES:
- [Background] Jadzinsky M, Pfutzner A, Paz-Pacheco E, Xu Z, Allen E, Chen R; CV181-039 Investigators. Saxagliptin given in combination with metformin as initial therapy improves glycaemic control in patients with type 2 diabetes compared with either monotherapy: a randomized controlled trial. Diabetes Obes Metab. 2009 Jun;11(6):611-22. doi: 10.1111/j.1463-1326.2009.01056.x. PMID 19515181
- [Derived] Gnesin F, Thuesen ACB, Kahler LKA, Madsbad S, Hemmingsen B. Metformin monotherapy for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Jun 5;6(6):CD012906. doi: 10.1002/14651858.CD012906.pub2. PMID 32501595
- [Derived] Cook W, Minervini G, Bryzinski B, Hirshberg B. Saxagliptin efficacy and safety in patients with type 2 diabetes mellitus stratified by cardiovascular disease history and cardiovascular risk factors: analysis of 3 clinical trials. Postgrad Med. 2014 Oct;126(6):19-32. doi: 10.3810/pgm.2014.10.2818. PMID 25414932
- [Derived] Karyekar CS, Frederich R, Ravichandran S. Clinically relevant reductions in HbA1c without hypoglycaemia: results across four studies of saxagliptin. Int J Clin Pract. 2013 Aug;67(8):759-67. doi: 10.1111/ijcp.12212. Epub 2013 Jun 24. PMID 23795975
- [Derived] Pfutzner A, Paz-Pacheco E, Allen E, Frederich R, Chen R; CV181039 Investigators. Initial combination therapy with saxagliptin and metformin provides sustained glycaemic control and is well tolerated for up to 76 weeks. Diabetes Obes Metab. 2011 Jun;13(6):567-76. doi: 10.1111/j.1463-1326.2011.01385.x. PMID 21342412

RESULTS

PARTICIPANT FLOW:
Groups:
- Saxagliptin 5 mg + Metformin: The Saxagliptin 5 mg + Metformin group includes data from participants randomized to receive coadministration of blinded, fixed-dose saxagliptin 5 mg oral tablets and metformin IR 500 mg. Metformin Immediate Release (IR) was titrated, as tolerated, in increments of 500 mg up to a maximum of 2000 mg daily dose.
- Saxagliptin 10 mg + Metformin: The Saxagliptin 10 mg + Metformin group includes data from participants randomized to receive coadministration of blinded, fixed-dose saxagliptin 10 mg oral tablets and metformin IR 500 mg. Metformin IR was titrated, as tolerated, in increments of 500 mg up to a maximum of 2000 mg daily dose.
- Saxagliptin 10 mg: The Saxagliptin 10 mg group includes data from participants randomized to receive coadministration of blinded, fixed-dose saxagliptin 10 mg oral tablets and placebo resembling metformin.
- Metformin: The Metformin group includes data from participants randomized to receive coadministration of metformin IR 500 mg. Metformin IR was titrated, as tolerated, in increments of 500 mg up to a maximum of 2000 mg daily dose and placebo resembling saxagliptin.
Period: Overall Study
Arm/Group | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Saxagliptin 10 mg | Metformin
Started | 320 | 323 | 335 | 328
Completed Study Without Being Rescued | 179 | 177 | 113 | 144
Completed | 229 | 231 | 209 | 219
Not Completed | 91 | 92 | 126 | 109
Not completed — Lack of Efficacy | 18 | 18 | 35 | 29
Not completed — Withdrawal of Consent by Subject | 20 | 24 | 28 | 25
Not completed — Lost to Follow-up | 22 | 23 | 29 | 22
Not completed — Adverse Event | 14 | 10 | 14 | 14
Not completed — Subject no longer meets study criteria | 4 | 2 | 8 | 7
Not completed — Poor/Noncompliance | 11 | 8 | 4 | 5
Not completed — Physician Decision | 0 | 1 | 3 | 2
Not completed — Death | 1 | 2 | 2 | 3
Not completed — Pregnancy | 0 | 2 | 1 | 1
Not completed — Administrative Reason by Sponsor | 1 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Saxagliptin 10 mg | Metformin | Total
Number analyzed (Participants) | 320 | 323 | 335 | 328 | 1306
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.95 (10.43) | 52.08 (11.59) | 52.09 (10.17) | 51.83 (10.74) | 51.99 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 177 | 166 | 165 | 663
  Male | 165 | 146 | 169 | 163 | 643

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (A1C) at Week 24, Saxagliptin Plus Metformin Versus Saxagliptin Monotherapy
Description: Mean change from baseline in A1C at Week 24, adjusted for baseline value.
Time Frame: Baseline, Week 24
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in analysis of change from baseline to Week 24 Last Observation Carried Forward (LOCF), subjects must have had a baseline and at least 1 post-baseline measurement. If participant received rescue medication, that measurement must have been taken before rescue.
Measure: Mean (Standard Error); unit: percent
Groups:
- Saxagliptin 5 mg + Metformin: The Saxagliptin 5 mg + Metformin group includes data from participants randomized to receive coadministration of blinded, fixed-dose saxagliptin 5 mg oral tablets and metformin IR 500 mg. Metformin IR was titrated, as tolerated, in increments of 500 mg up to a maximum of 2000 mg daily dose.
Arm/Group | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Saxagliptin 10 mg
Number analyzed (Participants) | 306 | 315 | 317
percent
  Baseline Mean | 9.41 (0.072) | 9.53 (0.069) | 9.61 (0.075)
  Week 24 Mean | 6.93 (0.066) | 7.02 (0.067) | 7.86 (0.085)
  Adjusted Mean Change from Baseline | -2.53 (0.070) | -2.49 (0.069) | -1.69 (0.069)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24, Saxagliptin Plus Metformin Versus Saxagliptin Monotherapy
Description: Mean change from baseline in FPG at Week 24, adjusted for baseline value.
Time Frame: Baseline, Week 24
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in analysis of change from baseline to Week 24 LOCF, participants must have had a baseline and at least 1 post-baseline measurement. If a participant received rescue medication, then that measurement must have been taken before rescue.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Saxagliptin 10 mg
Number analyzed (Participants) | 315 | 317 | 327
mg/dL
  Baseline Mean | 198.9 (3.17) | 204.3 (3.35) | 200.9 (3.03)
  Week 24 Mean | 140.2 (2.39) | 140.1 (2.34) | 169.9 (3.20)
  Adjusted Mean Change from Baseline | -59.8 (2.34) | -62.2 (2.34) | -30.9 (2.30)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24, Saxagliptin Plus Metformin Versus Metformin Monotherapy
Description: Mean change from baseline in FPG at Week 24, adjusted for baseline value.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Metformin
Number analyzed (Participants) | 315 | 317 | 320
mg/dL
  Baseline Mean | 198.9 (3.17) | 204.3 (3.35) | 199.1 (3.28)
  Week 24 Mean | 140.2 (2.39) | 140.1 (2.34) | 152.7 (2.80)
  Adjusted Mean Change from Baseline | -59.8 (2.34) | -62.2 (2.34) | -47.3 (2.33)

4. Secondary Outcome: Percentage of Participants Achieving A1C < 7% at Week 24, Saxagliptin Plus Metformin Versus Saxagliptin Monotherapy
Description: Percentage of participants achieving A1C < 7%, the American Diabetes Association's defined goal for glycemia, at each dose of saxagliptin plus metformin versus saxagliptin alone at Week 24.
Time Frame: Week 24
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in the Week 24 LOCF analysis, participants must have had at least 1 post-baseline measurement. If a participant received rescue medication, then that measurement must have been taken before rescue.
Measure: Number; unit: Percentage of participants
Arm/Group | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Saxagliptin 10 mg
Number analyzed (Participants) | 307 | 315 | 320
Percentage of participants | 60.3 | 59.7 | 32.2

5. Secondary Outcome: Percentage of Participants Achieving A1C < 7% at Week 24, Saxagliptin Plus Metformin Versus Metformin Monotherapy
Description: Percentage of participants achieving A1C < 7%, the American Diabetes Association's defined goal for glycemia, at each dose of saxagliptin plus metformin versus metformin alone at Week 24.
Time Frame: Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Metformin
Number analyzed (Participants) | 307 | 315 | 314
Percentage of participants | 60.3 | 59.7 | 41.1

6. Secondary Outcome: Changes From Baseline in Postprandial Glucose (PPG) Area Under the Curve (AUC) Response to an Oral Glucose Tolerance Test (OGTT) at Week 24, Saxagliptin Plus Metformin Versus Saxagliptin Monotherapy
Description: Mean change from baseline for 0 to 180 minutes PPG AUC at Week 24, adjusted for baseline value.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg*min/dL
Arm/Group | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Saxagliptin 10 mg
Number analyzed (Participants) | 142 | 131 | 145
mg*min/dL
  Baseline Mean | 55531 (1116.5) | 57219 (1169.6) | 57584 (1143.4)
  Week 24 Mean | 35324 (890.0) | 35790 (888.9) | 41229 (1050.9)
  Adjusted Mean Change from Baseline | -21080 (836.5) | -21336 (869.6) | -16054 (826.7)

7. Primary Outcome: Change From Baseline in A1C at Week 24, Saxagliptin Plus Metformin Versus Metformin Monotherapy
Description: Mean change from baseline in A1C at Week 24, adjusted for baseline value.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percent
Arm/Group | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Metformin
Number analyzed (Participants) | 306 | 315 | 313
percent
  Baseline Mean | 9.41 (0.072) | 9.53 (0.069) | 9.43 (0.073)
  Week 24 Mean | 6.93 (0.066) | 7.02 (0.067) | 7.48 (0.084)
  Adjusted Mean Change from Baseline | -2.53 (0.070) | -2.49 (0.069) | -1.99 (0.069)

8. Secondary Outcome: Changes From Baseline in Postprandial Glucose (PPG) Area Under the Curve (AUC) Response to an Oral Glucose Tolerance Test (OGTT) at Week 24, Saxagliptin Plus Metformin Versus Metformin Monotherapy
Description: Mean change from baseline for 0 to 180 minutes PPG AUC at Week 24, adjsuted for baseline value.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg*min/dL
Arm/Group | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Metformin
Number analyzed (Participants) | 142 | 131 | 135
mg*min/dL
  Baseline Mean | 55531 (1116.5) | 57219 (1169.6) | 57937 (1281.7)
  Week 24 Mean | 35324 (890.0) | 35790 (888.9) | 42428 (1082.1)
  Adjusted Mean Change from Baseline | -21080 (836.5) | -21336 (869.6) | -15005 (857.0)

9. Secondary Outcome: Percentage of Participants Achieving A1C ≤6.5% at Week 24, Saxagliptin Plus Metformin Versus Saxagliptin Monotherapy
Description: Percentage of participants achieving A1C ≤6.5%, at each dose of saxagliptin plus metformin versus saxagliptin alone at Week 24.
Time Frame: Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Saxagliptin 10 mg
Number analyzed (Participants) | 307 | 315 | 320
Percentage of Participants | 45.3 | 40.6 | 20.3

10. Secondary Outcome: Percentage of Participants Achieving A1C ≤6.5% at Week 24, Saxagliptin Plus Metformin Versus Metformin Monotherapy
Description: Percentage of participants achieving A1C ≤6.5%, at each dose of saxagliptin plus metformin versus metformin alone at Week 24.
Time Frame: Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Metformin
Number analyzed (Participants) | 307 | 315 | 314
Percentage of participants | 45.3 | 40.6 | 29.0

11. Secondary Outcome: Percentage of Participants Requiring Rescue or Discontinuation at Week 24, Saxagliptin Plus Metformin Versus Saxagliptin Monotherapy
Description: Percentage of participants requiring rescue for failing to achieve pre-specified glycemic targets or discontinuing for lack of efficacy within the 24-week treatment period at each dose of saxagliptin plus metformin versus saxagliptin alone.
Time Frame: Week 24
Population: Randomized participants who took at least 1 dose of double-blind treatment were included in the Week 24 LOCF analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Saxagliptin 10 mg
Number analyzed (Participants) | 320 | 323 | 335
Percentage of participants | 7.5 | 5.9 | 21.2

12. Secondary Outcome: Percentage of Participants Requiring Rescue or Discontinuation at Week 24, Saxagliptin Plus Metformin Versus Metformin Monotherapy
Description: Percentage of participants requiring rescue for failing to achieve pre-specified glycemic targets or discontinuing for lack of efficacy within the 24-week treatment period at each dose of saxagliptin plus metformin versus metformin alone.
Time Frame: Week 24
Population: Randomized participants who took at least 1 dose of double-blind treatment were included in the Week 24 LOCF analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Saxagliptin 5 mg + Metformin | Saxagliptin 10 mg + Metformin | Metformin
Number analyzed (Participants) | 320 | 323 | 328
Percentage of participants | 7.5 | 5.9 | 10.1

ADVERSE EVENTS:
Arm/Group | Metformin | Saxagliptin 10 mg | Saxagliptin 10 mg + Metformin | Saxagliptin 5 mg + Metformin
Serious Adverse Events (participants affected / at risk) | 15/328 | 16/335 | 22/323 | 16/320
Other Adverse Events (participants affected / at risk) | 106/328 | 106/335 | 122/323 | 116/320
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin (N=328) | Saxagliptin 10 mg (N=335) | Saxagliptin 10 mg + Metformin (N=323) | Saxagliptin 5 mg + Metformin (N=320)
DIABETIC RETINOPATHY (Eye disorders) | 0 | 1 | 0 | 0
CARDIAC ARREST (Cardiac disorders) | 0 | 0 | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 2 | 0 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 0 | 1 | 1
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 0 | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 2 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 0 | 0 | 1
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 | 1 | 0 | 0
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 0 | 1 | 0 | 0
EXTREMITY NECROSIS (Vascular disorders) | 0 | 0 | 1 | 0
DIABETIC MACROANGIOPATHY (Vascular disorders) | 0 | 1 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 1 | 0 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0 | 0 | 0
SCIATICA (Nervous system disorders) | 0 | 1 | 0 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 0 | 1 | 0 | 0
SYNCOPE VASOVAGAL (Nervous system disorders) | 1 | 0 | 0 | 0
CEREBRAL INFARCTION (Nervous system disorders) | 0 | 0 | 0 | 1
HAEMORRHAGIC STROKE (Nervous system disorders) | 0 | 0 | 1 | 0
FACIAL NERVE DISORDER (Nervous system disorders) | 0 | 0 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0 | 0 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 1
PANCREATITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
HIATUS HERNIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
FOOD POISONING (Gastrointestinal disorders) | 1 | 0 | 0 | 0
GASTRIC POLYPS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 | 0 | 1 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 0 | 1 | 0
DEAFNESS (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
SEPSIS (Infections and infestations) | 1 | 0 | 0 | 0
TETANUS (Infections and infestations) | 0 | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 1 | 0 | 0
ERYSIPELAS (Infections and infestations) | 0 | 0 | 0 | 1
APPENDICITIS (Infections and infestations) | 0 | 1 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 1
SCROTAL ABSCESS (Infections and infestations) | 0 | 0 | 1 | 0
PHARYNGOTONSILLITIS (Infections and infestations) | 0 | 0 | 1 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 1 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 0 | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
LYMPHADENITIS (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
ROSACEA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
MENOMETRORRHAGIA (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
ACQUIRED PHIMOSIS (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
ACCIDENT (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
PYREXIA (General disorders) | 0 | 0 | 1 | 0
SUDDEN DEATH (General disorders) | 1 | 0 | 1 | 0
PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
BILE DUCT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
LYMPHOPROLIFERATIVE DISORDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin (N=328) | Saxagliptin 10 mg (N=335) | Saxagliptin 10 mg + Metformin (N=323) | Saxagliptin 5 mg + Metformin (N=320)
HYPERTENSION (Vascular disorders) | 17 | 19 | 21 | 27
HEADACHE (Nervous system disorders) | 18 | 31 | 36 | 31
DIARRHOEA (Gastrointestinal disorders) | 30 | 12 | 41 | 26
INFLUENZA (Infections and infestations) | 19 | 17 | 13 | 20
NASOPHARYNGITIS (Infections and infestations) | 19 | 24 | 19 | 29
URINARY TRACT INFECTION (Infections and infestations) | 25 | 23 | 22 | 13
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 | 14 | 19 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.